CLINICAL TRIAL: NCT00176865
Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With Immunologic or Histiocytic Disorders Using a Non-Myeloablative Preparative Regimen to Achieve Stable Mixed Chimerism
Brief Title: Stem Cell Transplant for Immunologic or Histiocytic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2002-12; 0207M29448 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hemophagocytic Lymphohistiocytosis; X-Linked Lymphoproliferative Disorders; Chediak-Higashi Syndrome; Griscelli Syndrome; Immunologic Deficiency Syndromes; Langerhans-Cell Histiocytosis
Keywords: Stem cell transplant; immunodeficiency; donor lymphocyte infusion
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Lymphoproliferative Disorders; Chediak-Higashi Syndrome; Immunologic Deficiency Syndromes; Histiocytosis, Langerhans-Cell | interventions — Stem Cell Transplantation; fludarabine; fludarabine phosphate; Melphalan; Antilymphocyte Serum; Alemtuzumab; Cyclosporine; Mycophenolic Acid; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 - Matched sibling donor (Active Comparator): Stem Cell Transplant: human leukocyte antigen (HLA) genotypic matched sibling donor and pre-treatment with fludarabine, melphalan, anti-thymocyte globulin or Campath 1H and post-treatment with Cyclosporin A, mycophenolate mofetil and Intravenous immunoglobulin (IVIG)
  Interventions: Procedure: Stem Cell Transplant; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (ATG); Drug: Campath 1H; Drug: Cyclosporin A; Drug: Mycophenolate mofetil; Drug: Intravenous immunoglobulin (IVIG)
- Arm 2 - Matched unrelated donor (Active Comparator): Stem Cell Transplant: HLA phenotypic matched unrelated peripheral blood stem cell (PBSC) donor and pre-treatment with fludarabine, melphalan, anti-thymocyte globulin or Campath 1H and post-treatment with Cyclosporin A, mycophenolate mofetil and Intravenous immunoglobulin (IVIG)
  Interventions: Procedure: Stem Cell Transplant; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (ATG); Drug: Campath 1H; Drug: Cyclosporin A; Drug: Mycophenolate mofetil; Drug: Intravenous immunoglobulin (IVIG)
- Arm 3 - Mismatched double cord donors (Active Comparator): Stem Cell Transplant: two HLA 0-2 antigen mismatched unrelated cord blood donors (double cord) and pre-treatment with fludarabine, melphalan, anti-thymocyte globulin or Campath 1H and post-treatment with Cyclosporin A, mycophenolate mofetil and Intravenous immunoglobulin (IVIG)
  Interventions: Procedure: Stem Cell Transplant; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (ATG); Drug: Campath 1H; Drug: Cyclosporin A; Drug: Mycophenolate mofetil; Drug: Intravenous immunoglobulin (IVIG)

INTERVENTIONS:
Procedure: Stem Cell Transplant — IV on Day 0
  Other Names: hematopoietic stem cell transplant
Drug: Fludarabine — 30mg/m^2 IV Day -7 through Day -3
  Other Names: Fludara
Drug: Melphalan — 140 mg/m^2 IV Day -1
  Other Names: Alkeran
Drug: Anti-thymocyte globulin (ATG) — 30 mg/kg IV Day -5 through Day -1
  Other Names: ATGAM
Drug: Campath 1H — 0.2 mg/kg IV X 5 days (used as an alternative to Anti-thymocyte globulin (ATG) if unable to tolerate ATG) Day -10 through Day -6
  Other Names: Alemtuzumab
Drug: Cyclosporin A — 2.5 mg/kg IV every 12 hours (adults) or every 8 hours (children <40 kg) maintaining a level of >200mg/L Day -3 until Day +180 when, if no GVHD, the dose will be tapered 10% per week beginning on day 181
Drug: Mycophenolate mofetil — 15 mg/kg IV or orally bid and discontinued on Day +45 unless GVHD is present
  Other Names: CellCept
Drug: Intravenous immunoglobulin (IVIG) — 500 mg/kg IV weekly beginning on Day +7 until Day +100

SUMMARY:
This study tests the clinical outcomes of a preparative regimen of fludarabine (FLU), anti-thymocyte globulin (ATG)/or Campath, and melphalan; followed by hematopoietic stem cell transplant, and a post transplant regimen of Cyclosporin A (CsA) in patients with immunologic or histiocytic disorders. The researchers hypothesize that this regimen will have a positive effect on post transplant engraftment and the incidence of graft-versus-host-disease (GVHD).

Patients will be randomized biologically into one of 3 arms based upon donor availability: (a) human leukocyte antigen (HLA) genotypic matched sibling donor, (b) HLA phenotypic matched unrelated peripheral blood stem cell (PBSC) donor, (c) two HLA 0-2 antigen mismatched unrelated cord blood donors (double cord).

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive Melphalan, Fludarabine and Anti-Thymocyte Globulin (ATG) or Campath. These three drugs are being given to subjects to help the new stem cells take and grow. On the day of transplantation, subjects will receive stem cells transfused via intravenous (IV) catheter.

After stem cell transplantation, subjects will be given Cyclosporin A (CsA) and mycophenolate mofetil (MMF) to reduce the risk of graft-versus-host disease, the complication that occurs when the donor's stem cells react against the patient.

ELIGIBILITY:
Inclusion Criteria:

Patients with immunodeficiencies or histiocytic disorders 0-35 years of age with an acceptable stem cell donor and disease characteristic defined by the following:

* Patients with histocytic disorders (hemophagocytic lymphohistiocytosis of any etiology and refractory Langerhans cell histiocytosis) who do not meet eligibility criteria for a myeloablative transplant procedure
* Patients with immunodeficiency disorders in whom residual immune function may not require a fully myeloablative preparative regimen or patient is ineligible for standard myeloablative preparative regimen (any form of severe combined immunodeficiency [SCID], or other immunodeficiency with T cell defect)
* Patients with immunodeficiency disorders that have had poor outcome with myeloablative stem cell transplants (including, but not limited to, common variable immunodeficiency [CVID], Wiskott Aldrich Syndrome [WAS] if > 5 years of age, ataxia telangiectasia)
* Patients with immunodeficiencies or histocytic disorders that require a second stem cell transplant (SCT) for any reason

Exclusion Criteria:

* Karnofsky or Lansky performance score <70
* Glomerular filtration rate (GFR)<30% predicted
* Cardiac function <50% normal by echocardiogram
* Serum creatinine > 2x normal for age/weight
* Pregnant or lactating females
* Active serious infection that has not had an adequate course of therapy pre-SCT. Any patient with acquired immune deficiency syndrome (AIDS) or AIDS-related complex (ARC) or human immunodeficiency virus (HIV) seropositivity

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2002-08; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Matched Sibling Donor: human leukocyte antigen (HLA) genotypic matched sibling donor
  Stem Cell Transplant: Reduced intensity chemotherapy followed by infusion of hematopoietic stem cells
  Fludarabine, melphalan, ATG or Campath: all drugs are given intravenously (IV). Fludarabine x 5 days and melphalan x 1 day
- Arm 2 - Matched Unrelated Donor: HLA phenotypic matched unrelated peripheral blood stem cell (PBSC) donor,
  Stem Cell Transplant: Reduced intensity chemotherapy followed by infusion of hematopoietic stem cells
  Fludarabine, melphalan, ATG or Campath: all drugs are given intravenously (IV). Fludarabine x 5 days and melphalan x 1 day
- Arm 3 - Mismatched Double Cord Donors: two HLA 0-2 antigen mismatched unrelated cord blood donors (double cord).
  Stem Cell Transplant: Reduced intensity chemotherapy followed by infusion of hematopoietic stem cells
  Fludarabine, melphalan, ATG or Campath: all drugs are given intravenously (IV). Fludarabine x 5 days and melphalan x 1 day
Period: Overall Study
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Started | 3 | 10 | 6
Completed | 3 | 10 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors | Total
Number analyzed (Participants) | 3 | 10 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 10 | 6 | 19
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 2 | 7 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Mixed Chimerism
Description: >10% Donor Cells at Day 100
Time Frame: Day 100
Population: Arm 2: 2 of 10 patients not evaluable due to failure to return to clinic for the Day 100 evaluation.
  Arm 3: 2 of 6 patients not evaluable due to early death.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 8 | 4
participants | 3 | 8 | 4

2. Secondary Outcome: Percentage of Donor Chimerism at 100 Days
Description: The percent of recipient bone marrow and blood cells that are of donor origin.
Time Frame: Day 100
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 8 | 4
percentage of donor cells | 96.5 (6.0) | 75.5 (37.3) | 100 (0)

3. Secondary Outcome: Percentage of Donor Chimerism at 180 Days
Description: The percent of recipient bone marrow and blood cells that are of donor origin.
Time Frame: Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 8 | 4
percentage of donor cells | 88.9 (19.2) | 73.3 (41.7) | 90.5 (16.4)

4. Secondary Outcome: Percentage of Donor Chimerism at 365 Days
Description: The percent of recipient bone marrow and blood cells that are of donor origin.
Time Frame: Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 8 | 4
percentage of donor cells | 81.9 (31.4) | 78.6 (38.2) | 91.7 (13.5)

5. Secondary Outcome: Incidence of Grade 2-4 Acute Graft Versus Host Disease (aGVHD)
Description: Acute graft versus host disease (aGVHD) is a reaction occurring within the first 100 days after transplant where the T- cells of the donor graft attacks the recipient's (host's) skin, GI tract, liver and other organs. The severity of aGVHD is graded on a scale of 1 - 4 with the highest number representing the most severe disease.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 10 | 6
participants | 1 | 3 | 0

6. Secondary Outcome: Incidence of Grade 3-4 Acute Graft Versus Host Disease (aGVHD)
Description: as for outcome 5
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 10 | 6
participants | 1 | 1 | 0

7. Secondary Outcome: Incidence of Chronic Graft Versus Host Disease (cGVHD)
Description: Chronic graft versus host disease (cGVHD) is a reaction which typically develops 3 to 6 months after transplant where the T- cells of the donor graft attacks the recipient's (host's) skin, GI tract, liver and other organs.
Time Frame: 6 months and 1 year
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 10 | 6
participants | 1 | 0 | 0

8. Secondary Outcome: Number of Subjects Alive at 100 Days
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 10 | 6
participants | 3 | 8 | 4

9. Secondary Outcome: Number of Subjects Alive at One Year
Time Frame: Day 365
Measure: Number; unit: participants
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 3 | 10 | 6
participants | 3 | 7 | 3

10. Secondary Outcome: Compare Quality of Life (QOL)
Time Frame: Pretransplant, 1 year, 2 years and 5 years
Population: PI made decision after IRB approval, but before opening the study to accrual, to not collect QOL data .
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 - Matched Sibling Donor | Arm 2 - Matched Unrelated Donor | Arm 3 - Mismatched Double Cord Donors
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 2/3 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Matched Sibling Donor (N=3) | Arm 2 - Matched Unrelated Donor (N=10) | Arm 3 - Mismatched Double Cord Donors (N=6)
Multi-organ failure (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Matched Sibling Donor (N=3) | Arm 2 - Matched Unrelated Donor (N=10) | Arm 3 - Mismatched Double Cord Donors (N=6)
Hypertension (Cardiac disorders) | 1 | 4 | 1
Delayed growth (Endocrine disorders) | 1 | 2 | 0
Infection, GI (Infections and infestations) | 1 | 3 | 2
Cystitis (Renal and urinary disorders) | 1 | 2 | 0
Infection, blood (Infections and infestations) | 1 | 7 | 1
Delirious (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0
Incipient cataracts, bilateral (Eye disorders) | 1 | 0 | 0
Hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Infection, respiratory (Infections and infestations) | 1 | 8 | 5
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Infection, skin (Infections and infestations) | 1 | 0 | 0
Acute renal failure (Renal and urinary disorders) | 0 | 1 | 1
GI bleed (Gastrointestinal disorders) | 0 | 2 | 1
Capillary leak (Vascular disorders) | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Colonic pneumatosis (Gastrointestinal disorders) | 0 | 1 | 0
Erythrodermic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemorrhagic cystitis (Renal and urinary disorders) | 0 | 1 | 0
Hemorrhagic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Hyperbilirubinemia (Investigations) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
ICU dementia (Psychiatric disorders) | 0 | 1 | 0
Infection, GU (Infections and infestations) | 0 | 3 | 1
Liver failure (Hepatobiliary disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucositis (Gastrointestinal disorders) | 0 | 1 | 1
Otitis (Infections and infestations) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Prerenal azotemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Prolonged QTC interval (Cardiac disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1
Skin breakdown (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subclavian thrombosis (Vascular disorders) | 0 | 1 | 0
Veno-occlusive disease (Hepatobiliary disorders) | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Cholestasis portal fibrosis and bile duct proliferation (Hepatobiliary disorders) | 0 | 0 | 1
Ear drainage (Ear and labyrinth disorders) | 0 | 0 | 1
Elevated liver function tests (Investigations) | 0 | 0 | 1
Infection, NOS (Infections and infestations) | 0 | 0 | 1
Intraparenchymal hemorrhage, left frontal lobe (Nervous system disorders) | 0 | 0 | 1
Learning dysfunction (Nervous system disorders) | 0 | 0 | 1
Respiratory distress and apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Syndrome of inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No